CLINICAL TRIAL: NCT07333066
Title: Phase III Randomized International Open Label Clinical Trial of Treatment Intensification With Docetaxel Plus Apalutamide in Patients With Metastatic Hormone-sensitive Prostate Cancer Who Did Not Achieve a Deep PSA Response After Initial Treatment With Apalutamide: REINFORCE Trial.
Acronym: REINFORCE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alianza multidisciplinar para la investigación de los tumores genitourinarios -GUARD (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REINFORCE; 2025-524408-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer
Keywords: Prostate Cancer; Apalutamide; Hormone-sensitive prostate cancer; Deep PSA response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (experimental arm) (Experimental): Docetaxel (75 mg/m2 every three weeks), for 6 planned cycles, plus apalutamide (240 mg, oral single daily dose) and ADT.
  Interventions: Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets; Drug: Docetaxel
- Arm B (control arm) (No Intervention): Continuation of SOC treatment with apalutamide (240 mg, oral single daily dose) and ADT.

INTERVENTIONS:
Drug: Apalutamide (Erleada™) 60 mg or 240 mg tablets — The dose of 240 mg (four 60 mg tablets or one single 240 mg tablet) daily of apalutamide is the recommended dose in the SmPC.
  ADT will be chosen and administered according to standard clinical practice at each participating site and has not been included in the table below.
  Arms: Arm A (experimental arm)
Drug: Docetaxel — The recommended dose of docetaxel is 75 mg/m2 day 1 every 21 days. Six cycles of docetaxel will be administered.
  Arms: Arm A (experimental arm)

SUMMARY:
This is a phase III, randomized, open-label, multi-center study to assess the efficacy of treatment intensification with docetaxel plus apalutamide and ADT, assessed by event-free survival, in patients with mHSPC who do not achieve deep PSA response (≤0,2 ng/ml or PSA90 response in combination with a PSA ≤ 4 ng/ml) after initial treatment with apalutamide and ADT. A non-deep PSA response is defined as PSA > 0.2 ng/ml in combination with a PSA response < 90%, or a PSA response ≥90% in combination with a PSA > 4 ng/ml.

DETAILED DESCRIPTION:
Approximately 320 patients will be randomized in a 1:1 ratio to the treatments as specified below:

* Arm A (experimental arm): docetaxel (75 mg/m2 every three weeks), for 6 planned cycles, plus apalutamide and ADT (240 mg, oral single daily dose).
* Arm B (control arm): continuation of SOC treatment with apalutamide and ADT (240 mg, oral single daily dose).

Randomization will be stratified by 3 factors:

* Metastasis timing (synchronous vs metachronous)
* Visceral metastasis at diagnosis (yes vs no)
* PSA at study inclusion (≤ 4 ng/ml vs >4 ng/ml) An IDMC will be established for regular safety monitoring, for the pre-planned interim analysis and the PK sub-study when available. The composition, role, responsibilities and procedures of the IDMC will be detailed in the IDMC Charter.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent. Each patient must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures, required for the study, and is willing to participate in the study.
2. Patient must be a man ≥18 years of age.
3. Histologically or cytologically confirmed adenocarcinoma of prostate.
4. Metastatic hormone-sensitive prostate cancer.
5. PSA >5 ng/ml at diagnosis of metastatic disease.
6. Patients eligible to continue treatment with apalutamide and ADT and without contra-indication to receive docetaxel.
7. Patients with at least 24 weeks and no more than 30 weeks of apalutamide.
8. Patients with a maximum of 12 weeks ADT before apalutamide initiation.
9. Lack of achievement of deep PSA response after 24 weeks and no more than 30 weeks of apalutamide. Deep PSA response is defined as PSA ≤ 0.2 ng/ml or PSA response ≥ 90% in combination with a PSA ≤4 ng/ml. Therefore, a non-deep PSA response is defined as PSA > 0.2 ng/ml in combination with a PSA response < 90%, or a PSA response ≥90% in combination with a PSA > 4 ng/ml.
10. Patients who have not progressed to apalutamide.
11. Patients that are tolerating adequately apalutamide 240 mg daily and with no toxicity higher than G1 at inclusion.
12. Be able to swallow whole apalutamide film-coated tablets.
13. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
14. Clinical laboratory values at screening:

    1. hemoglobin ≥10.0 g/dL,
    2. absolute neutrophil count ≥1.5 × 10*9/L,
    3. platelet count ≥100 × 109/L, The patient must not have received any growth factor within 4 weeks or a blood transfusion within 7 days of the hematology laboratory sample obtained at screening
    4. serum alanine aminotransferase and/or aspartate transaminase ≤1.5 × the upper limit of normal (ULN),
    5. total bilirubin ≤ ULN,
    6. creatinine ≤2.0 × ULN
15. Sexually active men must agree to use an external condom as an effective barrier method and refrain from sperm donation, and their female partners of childbearing potential must practice a highly effective method of contraception during and for 3 months after treatment with apalutamide and for 6 months after treatment with docetaxel.

Exclusion Criteria:

1. Presence of neuroendocrine histology.
2. Apalutamide treatment started more than 30 weeks before inclusion.
3. Progression disease by any means, including radiographic, clinical or serological at inclusion.
4. Patient who achieves deep PSA response on apalutamide treatment before randomization.
5. Previous androgen-pathway receptor inhibitors, including enzalutamide, darolutamide, abiraterone or other ARPI. Previous treatment with first generation antiandrogens (i.e. bicalutamide) is allowed.
6. Chemotherapy or immunotherapy for prostate cancer before randomization.
7. Treatment with radiotherapy (external-beam radiation therapy, brachytherapy, or radiopharmaceuticals) within 2 weeks before randomization.
8. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs.
9. Contraindication to both computed tomography and magnetic resonance imaging contrast agent.
10. Any of the following within 6 months before randomization:

    1. stroke,
    2. myocardial infarction,
    3. severe or unstable angina pectoris,
    4. uncontrolled arrhythmia,
    5. coronary or peripheral artery bypass graft, or
    6. congestive heart failure (New York Heart Association class III or IV)
11. Peripheral neuropathy ≥ grade 2.
12. Uncontrolled hypertension, indicated by resting systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite medical management.
13. Prior malignancy, except for adequately treated basal-cell or squamous-cell carcinoma of the skin or superficial bladder cancer that had not spread behind the connective-tissue layer (i.e., stage pTis, pTa, or pT1) or any cancer for which treatment had been completed ≥5 years before randomization and from which the patient was disease-free.
14. A gastrointestinal disorder or procedure that was expected to interfere significantly with absorption of study drug.
15. Active viral hepatitis, known human immunodeficiency virus infection with detectable viral load, or chronic liver disease requiring treatment.
16. Previous (within 28 days before the start of study drug or 5 half-lives of the investigational treatment of the previous study, whichever was longer) or concomitant participation in another clinical study with investigational medicinal products.
17. Any other serious or unstable illness or medical, social, or psychological condition that could jeopardize the safety of the patient and/or their compliance with study procedures or might interfere with their participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | 48 months
  Event-free survival is defined as the time from randomization to occurrence of the following events, whichever occurs first in each treatment arm: PSA progression or radiographic progression of soft-tissue, visceral, or bone lesions or death from any cause.

SECONDARY OUTCOMES:
Time to castration resistance | 48 months
  Time to castration resistance is defined as time from randomization to radiographic disease progression, PSA progression per PCWG3 criteria, or symptomatic skeletal event (defined as radiation to bone, pathologic fracture, spinal cord compression, or surgery to bone due to symptoms), whichever occurred first in each treatment arm.
Radiographic progression-free survival (rPFS) | 48 months
  Radiographic Progression-Free Survival is defined as the time from randomization to the first documented evidence of radiographic disease progression, as assessed by the investigator per Prostate Cancer Working Group 3 (PCWG3) criteria for bone lesions and RECIST v1.1 for soft tissue lesions, or death from any cause, whichever occurs first in each treatment arm.
PSA progression-free survival | 48 months
  PSA progression-free survival (PSA-PFS) is defined according to PCWG3 criteria as the time from randomization to the date of PSA progression (a ≥25% increase and an absolute increase of ≥2 ng/mL from nadir, confirmed by a second value ≥3 weeks later) or death from any cause, whichever occurs first in each treatment arm.
Overall survival | 48 months
  Overall survival is defined as time from randomization to date of death from any cause in each treatment arm.
Time to subsequent treatment | 48 months
  Time to subsequent treatment is defined as the time from randomization to the initiation of the first subsequent systemic anticancer therapy after study drugs discontinuation, or death, whichever occurs first in each treatment arm.
Deep PSA response rate at 6 months in each treatment arm. | 6 months
  Deep PSA response is defined as achieving a prostate-specific antigen (PSA) level ≤0.2 ng/mL or PSA Response ≥90% in combination with a PSA ≤ 4 ng/ml.
Ultradeep PSA response rate at 6 months in each treatment arm. | 6 months
  Ultradeep PSA response 1 is defined as achieving a prostate-specific antigen (PSA) level between 0.2 and 0.02 ng/mL.
  Ultradeep PSA response 2 is defined as achieving a prostate-specific antigen (PSA) level ≤ 0.02 ng/mL.
Symptomatic skeletal event-free survival | 48 months
  Symptomatic skeletal event-free survival (SSE-FS) is defined as the time from randomization to the first occurrence of a symptomatic skeletal event (defined as radiation to bone, pathologic fracture, spinal cord compression, or surgery to bone due to symptoms) or death from any cause, whichever occurred first in each treatment arm.
To evaluate the safety profile of treatment intensification with docetaxel plus apalutamide and ADT (Adverse events) | 25 months
  Percentage of patients with at least one adverse event. Toxicity profile will be assessed using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0. Patients with each adverse event will be calculated over the total number of patients exposed in each treatment arm.
Time to initiate opioid use (≥ 7 days) | 48 months
  Time to initiate opioid use (≥ 7 days) is defined as the time from randomization to the first initiation of opioid analgesic use lasting for 7 or more consecutive days, regardless of the reason, or until death, whichever occurs first in each treatment arm.
To evaluate the safety profile of treatment intensification with docetaxel plus apalutamide and ADT (Serious adverse events). | 25 months
  Patients with at least a serious adverse event will be calculated over the total number of patients exposed in each treatment arm.
To evaluate the safety profile of treatment intensification with docetaxel plus apalutamide and ADT (Adverse events leading to treatment discontinuation ). | 25 months
  Patients with at least an adverse event leading to treatment discontinuation and adverse events leading to death will be calculated over the total number of patients exposed in each treatment arm.
To evaluate the safety profile of treatment intensification with docetaxel plus apalutamide and ADT (Death) | 25 months
  Dead patients calculated over the total number of patients exposed in each treatment arm.
To assess the quality of life of patients with FACT-P subscale | 24 months
  Change from baseline over time in FACT-P subscale in each treatment arm.
To assess the quality of life of patients with BPI-SF interference subscale | 24 months
  Change from baseline over time in BPI-SF interference subscale in each treatment arm.
To assess the quality of life of patients with BPI-SF interference subscale. | 24 months
  Change from baseline over time in BFI subscale in each treatment arm.

CONTACTS AND LOCATIONS:
Locations (56):
- France (20):
  - CH Bayonne, Bayonne
  - Institut Bergonié, Bordeaux
  - CHP Brest - Pasteur, Brest
  - Hôpital Henri-Mondor, Créteil
  - GHM Cancérologie - Institut Daniel Hollard, Grenoble
  - Hôpital Franco-Britannique, Levallois-Perret
  - GHBS - Hôpital du Scorff, Lorient
  - Centre De Cancérologie Du Grand Montpellier, Montpellier
  - Institut du Cancer de Montpellier - Val d'Aurelle (ICM), Montpellier
  - CHU Nîmes, Nîmes
  - Hospices Civils de Lyon - HCL, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Paris Saint-Joseph, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - Institut Godinot, Reims
  - CHU de Rennes, Rennes
  - Polyclinique Saint Georges, Saint-Georges-de-Didonne
  - CHP Saint Gregoire, Saint-Grégoire
  - Hôpital Foch, Suresnes
- Germany (9):
  - Facharztzentrum für Urologie, Uro-Onkologie, Berlin
  - Praxis Berlin / FASANUS - Urologie - Andrologie - Uro-Onkologie, Berlin
  - Johanniter-Krankenhaus Bonn-Gronau, Bonn
  - SRH Wald-Klinikum Gera, Gera
  - University Hospital Göttingen, Göttingen
  - Urologische Facharztpraxis Saale, Halle
  - Urologicum Karlsruhe MVZ, Karlsruhe
  - Klinikum Recklinghausen, Recklinghausen
  - University Hospital Rostock, Rostock
- Italy (5):
  - ARNAS Garibaldi - Catania, Catania
  - Hospital Riuniti di Foggia - Foggia, Foggia
  - National Instute of Oncology - Milan, Milan
  - Policlinico Gemelli Hospital - Rome, Roma
  - Policlinico Umberto I - Rome, Roma
- ULS Alto Ave, Guimarães, Portugal
- Spain (21):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitari Vall d´Hebron, Barcelona, Bacelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - ICO Badalona, Barcelona, Barcelona
  - Institut Català d'Oncologia (ICO) L´Hospitalet de Llobregat, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario 12 Octubre, Madrid, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Fundación Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid